CLINICAL TRIAL: NCT02311426
Title: Stroke in North of Norway and Denmark. A Prospective Cohort Study.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Audny Anke, MD, PhD, Professor, University Hospital of North Norway
Other Study IDs: SFP1175-14
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Stroke
Keywords: Rehabilitation; Functional outcome
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Norway: 500 consecutive patients with stroke from the stroke units at the University Hospital of North Norway located in the cities Narvik, Harstad and Tromsø.
  At baseline 155 patients with first ever stroke were registered. At 3 and 12 months follow-up 135-155 patients were enrolled.
  Interventions: Other: Observational study
- Denmark: 500 consecutive patients from the stroke unit at Århus Hospital in Denmark. At baseline 402 patients with first ever stroke were included. At 3 and 12 months follow-up 318/ 170 patients were enrolled.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Function, health related quality of life and rehabilitation needs will be analysed in the two country region groups

SUMMARY:
The study is a comparative effectiveness study with comparision of two cohorts of patients with stroke in North of Norway and in Denmark. At baseline information is collected from the stroke registries in both countries. Time points for follow up are at 3 and 12 months post-stroke. Data are collected from medical charts and with use of telephone interview in addition to self-report questionnaires. The study will provide information about functional status, health related quality of life and rehabilitation needs. Information about rehabilitation services in both countries are collected and compared, and analysed in relation to patients outcome.

ELIGIBILITY:
Inclusion Criteria:

* Verified stroke. Admitted to stroke unit.

Exclusion Criteria:

* Patients outside the regions excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke admitted to the stroke units at the University Hospital of North Norway and Århus Hospital in Denmark
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-03; Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Rehabilitation Needs | 3 months post-stroke
  Not enough help or training
Health related Quality of life questionnaire | 3 and 12 months post-stroke
  Qolibri_OS

CONTACTS AND LOCATIONS:
Overall Officials: Audny Anke, MD PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway